CLINICAL TRIAL: NCT03519009
Title: A Therapeutic Workplace to Address Poverty and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00160297; R01AA024101 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Substance Use Disorders
Keywords: Employment
MeSH Terms: conditions — Substance-Related Disorders | interventions — Myo-Inositol-1-Phosphate Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPS Plus Abstinence-Contingent Wage Supplement (Experimental): Abstinence-contingent wage supplements are provided for obtaining and maintaining competitive employment.
  Interventions: Behavioral: IPS Plus Abstinence-Contingent Wage Supplement
- Usual Care Control (No Intervention): Counseling and referrals to employment and treatment programs.

INTERVENTIONS:
Behavioral: IPS Plus Abstinence-Contingent Wage Supplement — Participants are offered abstinence-contingent wage supplements if they obtain and maintain competitive employment. The wage supplements are designed to promote employment while reinforcing drug abstinence. To help participants obtain and maintain competitive employment, participants will receive Individual Placement and Support (IPS) supported employment. IPS is a supported employment intervention that has been proven effective in promoting employment in adults with severe mental illness. To promote employment and prevent relapse to drug use, participants will receive IPS Plus Abstinence-Contingent Wage Supplements.
  Arms: IPS Plus Abstinence-Contingent Wage Supplement

SUMMARY:
Addiction is a chronic relapsing disorder. High magnitude and long-duration voucher-based abstinence reinforcement is one of the most effective treatments for alcohol and drug addiction and can maintain abstinence over extended periods of time, but practical methods of implementing these interventions are needed. Workplaces could be ideal and practical vehicles for arranging and maintaining abstinence reinforcement over long time periods. Investigators' research on a model Therapeutic Workplace has shown that employment-based abstinence reinforcement, in which participants must provide alcohol- or drug-free urine samples to maintain maximum pay, can maintain alcohol and drug abstinence. Now investigators need to develop effective and economically sound methods to arrange long-term exposure to employment-based abstinence reinforcement. Investigators are proposing to evaluate the effectiveness and economic benefits of a Wage Supplement Model of arranging long-term exposure to employment-based abstinence reinforcement. Under this model, successful Therapeutic Workplace participants are offered abstinence-contingent wage supplements if they obtain and maintain competitive employment. Governments have used wage supplements effectively to increase employment in welfare recipients. The Wage Supplement Model harnesses the power of wage supplements to promote employment, while simultaneously using the wage supplements to reinforce drug and alcohol abstinence. The intervention will combine 3 elements -- the Therapeutic Workplace, Individual Placement and Support (IPS) supported employment, and abstinence-contingent wage supplements. IPS is a supported employment intervention that has been proven effective in promoting employment in adults with severe mental illness. Under this model, participants will be exposed to the Therapeutic Workplace to initiate abstinence and establish job skills. To promote employment and prevent relapse to drug use, participants will receive IPS Plus Abstinence-Contingent Wage Supplements. A randomized trial will evaluate the effectiveness and economic benefits of the Abstinence-Contingent Wage Supplement Model in promoting employment and sustaining drug abstinence. Participants will be enrolled in the Therapeutic Workplace for 3 months and then randomly assigned to a Usual Care Control group or an IPS Plus Abstinence-Contingent Wage Supplement group for one year. Usual Care Control participants will be offered counseling and referrals to employment and treatment programs. IPS Plus Abstinence-Contingent Wage Supplement participants will receive the IPS intervention and abstinence-contingent wage supplements. This novel intervention could be an effective and economically sound way to promote long-term employment and drug abstinence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* meet Diagnostic and Statistical Manual (DSM-V) criteria for substance use disorder
* interested in obtaining employment

Exclusion Criteria:

* suicidal or homicidal ideation
* meet Diagnostic and Statistical Manual (DSM-V) criteria for psychotic disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novak MD, Toegel F, Holtyn AF, Rodewald AM, Arellano M, Baranski M, Barnett NP, Leoutsakos JM, Fingerhood M, Silverman K. Abstinence-contingent wage supplements for adults experiencing homelessness and alcohol use disorder: A randomized clinical trial. Prev Med. 2023 Nov;176:107655. doi: 10.1016/j.ypmed.2023.107655. Epub 2023 Aug 3. PMID 37541600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from treatment clinics and recovery houses serving adults with alcohol use disorder, online job boards, and through compensated referrals by participants. Participants were recruited from 2 January 2019 through 5 March 2020 and from 29 October 2020 through 12 May 2022. The pause in recruitment was due to regional and institutional restrictions related to the COVID-19 pandemic. Most of the study was conducted remotely because of the COVID-19 pandemic.
Pre-assignment Details: This was a two-group randomized clinical trial. All participants completed a 1-month Phase 1 Induction and Initiation period and were then randomly assigned to an intervention or control group. After random assignment, participants completed a 6-month Phase 2 Intervention period and completed study assessments every month.
Groups:
- Induction Period: During the first week, participants were introduced to the workplace contingencies: they could earn $5 per hour for up to 4 h per day for contacting research staff each day. Participants who contacted research staff 4 out of 5 days during the first week were invited to continue. During the next 3 weeks, participants were given a TAC monitoring device and could earn $8 per hour for up to 4 h per day each weekday. These devices had different requirements for use, which made it necessary for the procedures to be tailored to the device used. The SCRAM device requires that participants provide an alcohol-negative breath sample prior to use. Because participants had to be abstinent from alcohol to begin using SCRAM, participants fitted with SCRAM devices could maintain maximum pay if they continued abstaining from alcohol use. If alcohol use was detected, pay was reset to $1 per hour. After being reset, pay rates could be raised by $1 per hour (up to $8 per hour) for each day without alcohol use. The BACtrack Skyn device does not require that participants provide an alcohol-negative breath sample to begin using the device. So, incentives for alcohol abstinence were not provided during the Induction period for participants fitted with BACtrack Skyn. Instead, incentives were provided for wearing the device each day.
Period: Period 1, Phase 1
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control | Induction Period
Started | 0 | 0 | 152
Completed | 0 | 0 | 119
Not Completed | 0 | 0 | 33
Period: Period 2, Phase 2
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control | Induction Period
Started | 62 | 57 | 0
Completed | 62 | 57 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only randomized participants were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control | Total
Number analyzed (Participants) | 62 | 57 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (7.7) | 39.6 (8.5) | 39.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 52 | 49 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 19 | 24 | 43
  White | 42 | 31 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 57 | 119

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Abstinence
Description: Percentage of participants abstinent per month
Time Frame: 1 year
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control
Number analyzed (Participants) | 62 | 57
percentage of participants | 82.8 | 60.2
Statistical Analysis 1: Comparison: IPS Plus Abstinence-Contingent Wage Supplement vs Usual Care Control; Test type: Superiority; p < 0.001, longitudinal logistic regression; Odds Ratio (OR) = 3.4, 95% CI 2-sided [1.8 to 6.3]

2. Secondary Outcome: Employment
Description: Percentage of participants employed per month
Time Frame: 1 year
Population: intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control
Number analyzed (Participants) | 62 | 57
percentage of participants | 51.3 | 31.6
Statistical Analysis 1: Comparison: IPS Plus Abstinence-Contingent Wage Supplement vs Usual Care Control; Test type: Superiority; p < 0.001, longitudinal logistic regression; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.5 to 4.4]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | IPS Plus Abstinence-Contingent Wage Supplement | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/62 | 3/57
Other Adverse Events (participants affected / at risk) | 0/62 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPS Plus Abstinence-Contingent Wage Supplement (N=62) | Usual Care Control (N=57)
Hospitalization (General disorders) | 2 (2) | 3 (3)
Cancer (General disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03519009/Prot_SAP_000.pdf